CLINICAL TRIAL: NCT03375762
Title: REMOTE Ischemic Perconditioning Among Acute Ischemic Stroke Patients in CATalonia: REMOTE-CAT PROJECT
Brief Title: REMOTE Ischemic Perconditioning Among Acute Ischemic Stroke Patients ( REMOTE-CAT)
Acronym: REMOTE-CAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut de Recerca Biomèdica de Lleida (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Francisco Purroy, Professor. PHD. MD. Principal investigator of Neuroclinical sciences group, Institut de Recerca Biomèdica de Lleida
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: CEIC-1744
Record Dates: First submitted 2017-12-04; First posted 2017-12-18 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care plus RIPerC (Experimental): Usual care for stroke code patients, with or without revascularization therapies, with Remote ischemic perconditioning (RIPerC) using an electronic tourniquet.
  Interventions: Other: Remote ischemic perconditioning
- Usual care plus Sham RIPerC (Sham Comparator): Usual care for stroke code patients, with or without revascularization therapies, with Sham remote ischemic conditioning (RIPerC)
  Interventions: Other: Sham remote perconditioning

INTERVENTIONS:
Other: Remote ischemic perconditioning — Five 5-minute inflations/deflations of an automatic device placed on the upper non-paretic arm initiated in the ambulance on the way to hospital in the case of stroke code activation and RACE score >0 and RACE motor item>0
  Arms: Usual care plus RIPerC
Other: Sham remote perconditioning — Sham five 5-minute inflations/deflations of an automatic device placed on the upper non-paretic arm initiated in the ambulance on the way to hospital in the case of stroke code activation and RACE score >0 and RACE motor item>0
  Arms: Usual care plus Sham RIPerC

SUMMARY:
Stroke is one of the leading causes of death worldwide and the main cause of incapacity. Currently, the only therapies for acute ischemic stroke (AIS) patients are the administration of recombinant tissue plasminogen activator (rt-PA) and/or endovascular treatment. Unfortunately, many patients cannot benefit from these therapies due to contraindications or evolution time. Neuroprotective therapies could not only increase the benefits of available reperfusion therapies but also provide an option for patients who are not candidates for these treatments. Remote ischemic conditioning, consisting on brief episodes of transient limb ischemia, represents a new paradigm in neuroprotection. It can be categorized in pre-, per- or postconditioning, depending on the moment of application. According to studies in coronary ischemia, remote ischemic perconditioning (RIPerC) during the ischemic event is safe, cost-effective, feasible and associated with a reduction in myocardial injury. The investigators aim to conduct a multicentre study (5 university hospitals) of pre-hospital RIPerC in AIS patients (within 8 hours of stroke onset), which would include 572 stroke code activated patients (286 would undergo RIPerC and 286 would be sham). Our hypothesis is that RIPerC would be safe and would induce endogenous neuroprotective phenomena associated with good outcomes in AIS patients whether treated with revascularization therapies or not. Moreover, the development of systemic ischemic tolerance should provide metabolomic and lipidomic signatures that would present an opportunity to find specific molecular markers (biomarkers). The main objectives will be to assess: 1) RIPerC clinical benefits in AIS, 2) whether RIPerC is safe not only in AIS but also in all cases of stroke code activation, 3) whether RIPerC is associated with a reduction in cerebral infarct size and 4) metabolomic and lipidomic signatures of the RIPerC effect.

DETAILED DESCRIPTION:
Stroke is one of the leading causes of death worldwide and the main cause of incapacity. Currently, the only therapies for acute ischemic stroke (AIS) patients are the administration of rt-PA and/or endovascular treatment. Unfortunately, many patients cannot benefit from these therapies due to contraindications or evolution time. Neuroprotective therapies could not only increase the benefits of available reperfusion therapies but also provide an option for patients who are not candidates for these treatments. However, most neuroprotection trials have so far failed to demonstrate their efficacy in acute phase stroke patients, despite good results in animal studies. Remote ischemic perconditioning (RIPerC) represents a new paradigm in neuroprotection. It upregulates endogenous defense systems to achieve ischemic tolerance in brain ischemia. It consists of brief episodes of transient limb ischemia. According to studies in coronary ischemia, RIPerC during the ischemic event is safe, feasible and related to reduction in myocardial injury. However, there is only limited data about the clinical utility of RIC in AIS patients. Only one small single-centre, randomized, open label clinical trial has been conducted to test RIPerC in AIS patients as an adjunctive therapy intravenous alteplase in the prehospital setting.

The investigators want to conduct a multicenter study (involving 5 university hospitals) of prehospital RIPerC in AIS patients (within 8 hours of stroke onset) in which 572 stroke code activated patients will be included (286 subjects will undergo RIPerC and 286 subjects will be sham). RIPerC will consist of five cycles of electronic tourniquet inflation during five minutes and deflation during five minutes. The main endpoint will be a good clinical outcome measured by the modified Rankin score. The investigators will also establish a secondary neuroimaging endpoint defined by the infarct size observed in a Magnetic resonance imaging performed at three days. In addition, the investigators will conduct a substudy of biomarkers in 100 patients.

Our hypothesis is that RIPerC will be safe and will induce endogenous neuroprotective phenomenon responsible for good outcome in AIS patients whether treated with revascularization therapies or not. Moreover, the development of systemic ischemic tolerance will provide a metabolomic and lipidomic signature that will offer the opportunity to find specific molecular markers (biomarkers).

Project Objectives:

* To assess RIPerC clinical benefit in AIS measured by the modified Rankin Scale (mRS) score <3.
* To evaluate whether RIPerC is safe not only in AIS but also in all cases of stroke code activation.
* To assess whether RIPerC is associated with a reduction of cerebral infarct size.
* To identify the metabolomic and lipidomic signatures of the RIPerC effect.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years old
* Suspected clinical stroke with 8 hours since onset of neurological symptoms
* Stroke code (SC) activation
* Independent in daily life before the onset of acute symptoms. (mrs</=2)
* Rapid arterial occlusion evaluation (RACE) scale score>0 and RACE motor item>0
* Written informed consent (patient or representative)

Exclusion Criteria:

* Unknown onset of symptoms
* Coma (GCS< 8)
* Malignancy or significant co-morbidity thought to limit life expectancy to <6 months
* Pregnancy
* Taking part in another interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 572 (Estimated)
Dates: Start 2019-08-07 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Dependency | Day 90±7
  Modified Rankin Scale (MRS) <3. The mRS is an ordinal, graded interval scale that assigns patients among 7 global disability levels: 0 (no symptom) to 5 (severe disability) and 6 (death).

SECONDARY OUTCOMES:
Early neurological improvement rate | Day 1, day 5±1
  NIHSS decrease >=4 with respect to baseline
Treatment Related Serious Adverse Event Rates | Day 1, day 5±1, day 90±7
  Number of participants with a serious adverse event related to treatment
Size of the infarct volume | Day 5±1
  The infarct volume will be defined as the hyperintense area on the initial isotropic DWI acquired with a b value of 1000 sec/mm2
Symptomatic intracranial hemorrhage | 24-36 hours
  Symptomatic intracerebral hemorrhage (SICH) defined by the Safe Implementation of Thrombolysis in Stroke Monitoring Study protocol
Omic's response | Day 1, day 3, day 5±1
  Metabolomic and lipidomic analyses to define a panel of serum biomarkers accurately related to Remote ischemic conditioning phenomenon.
Early dependency | Day 5±1,
  Modified Rankin Scale <3. The mRS is an ordinal, graded interval scale that assigns patients among 7 global disability levels: 0 (no symptom) to 5 (severe disability) and 6 (death).

CONTACTS AND LOCATIONS:
Locations (1):
- Biomedical Research Institute of Lleida (IRBLleida) Institut de Recerca Biomèdica de Lleida, Lleida, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hougaard KD, Hjort N, Zeidler D, Sorensen L, Norgaard A, Hansen TM, von Weitzel-Mudersbach P, Simonsen CZ, Damgaard D, Gottrup H, Svendsen K, Rasmussen PV, Ribe LR, Mikkelsen IK, Nagenthiraja K, Cho TH, Redington AN, Botker HE, Ostergaard L, Mouridsen K, Andersen G. Remote ischemic perconditioning as an adjunct therapy to thrombolysis in patients with acute ischemic stroke: a randomized trial. Stroke. 2014 Jan;45(1):159-67. doi: 10.1161/STROKEAHA.113.001346. Epub 2013 Nov 7. PMID 24203849
- [Background] England TJ, Hedstrom A, O'Sullivan S, Donnelly R, Barrett DA, Sarmad S, Sprigg N, Bath PM. RECAST (Remote Ischemic Conditioning After Stroke Trial): A Pilot Randomized Placebo Controlled Phase II Trial in Acute Ischemic Stroke. Stroke. 2017 May;48(5):1412-1415. doi: 10.1161/STROKEAHA.116.016429. Epub 2017 Mar 6. PMID 28265014
- [Background] Heusch G, Botker HE, Przyklenk K, Redington A, Yellon D. Remote ischemic conditioning. J Am Coll Cardiol. 2015 Jan 20;65(2):177-95. doi: 10.1016/j.jacc.2014.10.031. PMID 25593060
- [Background] Hess DC, Blauenfeldt RA, Andersen G, Hougaard KD, Hoda MN, Ding Y, Ji X. Remote ischaemic conditioning-a new paradigm of self-protection in the brain. Nat Rev Neurol. 2015 Dec;11(12):698-710. doi: 10.1038/nrneurol.2015.223. Epub 2015 Nov 20. PMID 26585977
- [Background] Pan J, Li X, Peng Y. Remote ischemic conditioning for acute ischemic stroke: dawn in the darkness. Rev Neurosci. 2016 Jul 1;27(5):501-10. doi: 10.1515/revneuro-2015-0043. PMID 26812782
- [Derived] Purroy F, Arque G, Jimenez-Fabrega X, Subirats T, Ropero JR, Vicente-Pascual M, Cardona P, Gomez-Choco M, Pagola J, Abilleira S, Rovira A, Cirer-Sastre R, Mauri-Capdevila G; REMOTE-CAT Trial Investigators. Prehospital application of remote ischaemic perconditioning in acute ischaemic stroke patients in Catalonia: the REMOTE-CAT clinical trial. EClinicalMedicine. 2025 Apr 25;83:103208. doi: 10.1016/j.eclinm.2025.103208. eCollection 2025 May. PMID 40337071
- [Derived] Purroy F, Arque G, Mauri G, Garcia-Vazquez C, Vicente-Pascual M, Pereira C, Vazquez-Justes D, Torres-Querol C, Vena A, Abilleira S, Cardona P, Forne C, Jimenez-Fabrega X, Pagola J, Portero-Otin M, Rodriguez-Campello A, Rovira A, Marti-Fabregas J. REMOTE Ischemic Perconditioning Among Acute Ischemic Stroke Patients in Catalonia: REMOTE-CAT PROJECT. Front Neurol. 2020 Sep 25;11:569696. doi: 10.3389/fneur.2020.569696. eCollection 2020. PMID 33101178